CLINICAL TRIAL: NCT05191472
Title: Phase II Study of Pembrolizumab in Multiple Myeloma Patients Relapsing After or Refractory to Anti-BCMA CAR-T Therapies
Brief Title: Pembrolizumab for the Treatment of Relapsed or Refractory Multiple Myeloma After Anti-BCMA CAR-T Therapies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Alfred Chung, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Alfred Chung, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212530; NCI-2021-13897 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-01-02; First posted 2022-01-13 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
Keywords: CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475

SUMMARY:
This phase II trial tests whether pembrolizumab works to shrink tumors in patients with multiple myeloma whose cancer has come back (relapsed) or did not respond to previous treatment (refractory) with anti-BCMA CAR-T therapies. Immunotherapy with pembrolizumab, may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate (ORR) of pembrolizumab in patients with relapsed or refractory multiple myeloma (MM) (RRMM) after anti-B-cell receptor maturation antigen (BCMA) chimeric antigen receptor T-cell (CAR-T) therapies.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of pembrolizumab in participants who relapsed or were refractory to anti-BCMA CAR-T therapies.

II. To evaluate the depth of response for patients treated with pembrolizumab who had previously relapsed after or were refractory to anti-BCMA CAR-T therapies.

III. To evaluate time-to-event outcomes, including time-to-next treatment (TNT), progression-free survival (PFS), and overall survival (OS) after initiation of pembrolizumab therapy.

EXPLORATORY OBJECTIVE:

I. To explore the immune profile after pembrolizumab treatment, including changes in absolute lymphocyte count (ALC) and lymphocyte subsets by flow-cytometry.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Participants will be followed for at least 30 days after last treatment or removal from study, or until death. Participants who have completed 35 cycles of therapy or discontinued treatment for reasons other than disease progression will be followed for up to 1-year, until removal from study, start of new anti-cancer therapy, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are 18 years of age or older on the day of signing informed consent with histologically confirmed diagnosis of multiple myeloma will be enrolled in this study.
2. Ability to understand a written informed consent document, and the willingness to sign it or a legally acceptable representative (if applicable).
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%). Evaluation of ECOG is to be performed within 7 days prior to the start of study treatment.
4. The effects of pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception for the duration of study participation and 120 days after last administration of study treatment.

   * Female participants are eligible if not pregnant, not breastfeeding, and one of the following:

     * Not a woman of childbearing potential (WOCBP) OR
     * WOCBP who agrees to follow contraceptive guidance during treatment period and at least 120 days following last dose of study treatment.
   * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 120 days after last administration of study treatment. Men should also refrain from donating sperm during this period.
5. Participants must have either

   * progressive disease after prior anti-BCMA CAR-T therapy and have not started another systemic anti-cancer therapy following progression after anti-BCMA CAR-T therapy. Patients who received localized radiotherapy alone for symptomatic relief of progressive disease following anti-BCMA CAR-T will be allowed.
   * OR
   * b. stable disease as best hematologic response after at least 30 days post anti-BCMA CAR-T infusion.

   Progression after anti-BCMA CAR-T is defined by International Myeloma Working Group (IMWG) criteria:
   1. Increase of > 25% from lowest response value in any one or more of the following:

      * Serum M-component and/or (the absolute increase must be > 0.5 g/dL).
      * Urine M-component and/or (the absolute increase must be > 200 mg/24 h).
      * Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved free light chain (FLC) levels. The absolute increase must be > 10 mg/dL.
      * Bone marrow plasma cell percentage: the absolute percentage must be > 10%.
   2. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas and/or
   3. Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
6. Time from date of anti-BCMA CAR-T infusion to date of first administration of pembrolizumab (study drug) must be ≥ 30 days. In order to be eligible for this study, participants must not be candidates for treatment regimens known to provide clinical benefit in MM as assessed by the treating physician and must have previously received or are intolerant to a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 antibody.
7. Diagnosis of symptomatic multiple myeloma defined as: clonal bone marrow plasma cells > 10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following calcium elevation, renal insufficiency, anemia, and bone abnormalities (CRAB) features and myeloma-defining events.

   1. Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL).
   2. Renal insufficiency: creatinine clearance < 40 mL per minute or serum creatinine > 177 micromol/L (> 2 mg/dL).
   3. Anemia: hemoglobin value of >20g/L below the lowest limit of normal, or a hemoglobin value <100 g/L.
   4. Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)/CT. If bone marrow has < 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement.
   5. Any one or more of the following biomarkers of malignancy:

      * 60% or greater clonal plasma cells on bone marrow examination.
      * Serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100 mg/L.
      * More than one focal lesion on magnetic resonance imaging (MRI) that is at least 5mm or greater in size.
8. Active and measurable disease, defined by serum paraprotein (M-protein) >= 0.5 g/dL, 24-hour urine Bence Jones protein of >= 200 mg, or abnormal serum free light chain ratio with involved light chain of >= 10 mg/dL (100 mg/L).
9. Have adequate organ function as defined below. Specimens must be collected within 10 days prior to the start of study treatment:

   1. Absolute neutrophil count (ANC) >= 500/microliter (uL) (within 10 days prior to the start of study treatment).
   2. Platelets >= 25 000/uL (within 10 days prior to the start of study treatment).
   3. Hemoglobin >= 8.0 g/dL (within 10 days prior to the start of study treatment).

      * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed.
      * No lower limit if cytopenia is related to bone marrow involvement.
   4. Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of study treatment).

      * Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl.
      * Creatinine clearance (CrCl) should be calculated per institutional standard.
   5. Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of study treatment).
   6. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (within 10 days prior to the start of study treatment).

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to study treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   * Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-programmed cell death protein 1 (anti PD-1), anti-programmed death-ligand 1 (anti PD-L1), or anti programmed cell death 1 ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX 40, Cluster of Differentiation 137 (CD137)).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study treatment initiation.

   1. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible.
   2. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received anti-BCMA CAR-T infusion < 30 days prior to study treatment initiation.
5. Has received subsequent systemic anti-cancer therapy following anti-BCMA CAR-T therapy. Participants who received localized radiotherapy alone for symptom control following anti-BCMA CAR-T therapy will be allowed to participate.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines are generally Messenger RNA (mRNA)-based or viral vector vaccines (replication-incompetent) and are allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

   * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
8. Has a diagnosis of primary immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Has an active history of a second malignancy requiring treatment, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Participants with the following low-risk or non-invasive malignancies will be allowed:

   1. Basal cell carcinoma of the skin.
   2. Squamous cell carcinoma of the skin.
   3. Carcinoma in-situ of the cervix.
   4. Carcinoma in-situ of the breast.
   5. Superficial bladder cancer.
   6. Incidental histologic finding of prostate cancer (T1a or T1b using the Classification of Malignant Tumors (TNM) [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative or considered very-low or low risk in which observation is reasonable.
   7. Other in-situ cancers. * Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
11. Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
14. Has an active infection requiring systemic therapy. Prophylactic antibiotics/antivirals are allowed.
15. Has a known history of human immunodeficiency virus (HIV) infection.
16. Has known active Hepatitis B virus infection (defined as Hepatitis B (HBV) deoxyribonucleic acid (DNA) detected or Hepatitis B surface antigen (HbsAg) positive) or known active Hepatitis C virus infection (defined as Hepatitis C (HCV) ribonucleic acid (RNA) qualitative detected). Subjects who have been vaccinated against hepatitis B (positive for hepatitis B surface antibody (HBsAB)) who are negative for other markers of prior hepatitis B infection (e.g., Hepatitis B core antibody (HBcAb) negative) are eligible. Subjects with past exposure or known history of hepatitis B infection (e.g., HBcAb positive) are eligible for the study provided that they are negative by assessment for HBV DNA and HbsAg. Subjects with a history of hepatitis C infection (defined as detectable HCV antibody) are eligible as long as they have a negative HCV viral load.
17. Has a known history of active Bacillus Tuberculosis (TB).
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had a history of allogenic bone marrow/tissue/solid organ transplant.
22. Has unmeasurable disease by serum/urine testing (oligo-secretory or non-secretory multiple myeloma).
23. Has diagnosis of Waldenstrom's disease, light chain amyloidosis, or polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes (POEMS) disease.
24. ECOG performance status >= 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Chung, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab): Participants received pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 1
  60-69 years | 1
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The International Myeloma Working Group (IMWG) uniform response criteria will be used to assess disease response and progression. The response rate is defined as the proportion of patients achieving a partial response (PR), very good partial response (VGPR), complete response (CR), or a stringent complete response (sCR) after 4 cycles of pembrolizumab therapy. A 95% confidence interval will also be reported.
Time Frame: Up to 4 cycles (1 cycle is equal to 21 days)
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Participants With Reported Treatment-related Adverse Events
Description: The safety population will consist of all participants who receive any amount of study treatment. Safety will be assessed by evaluation of AEs using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Specific AEs will be counted once for each participant for calculating rates but will be presented in total in participant listings including frequency of non-hematologic grade 3 or higher adverse events.
Time Frame: Up to 30 days after discontinuing study treatment, approximately 1 year and 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Proportion of Participants With Cytokine Release Syndrome (CRS)
Description: Proportion of participants with reported CRS as defined by the American Society for Transplantation and Cellular Therapy (ASTCT) will be reported.
Time Frame: Up to 30 days after discontinuing study treatment, approximately 1 year and 8 months
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Participants With Immune-effector Cell-associated Neurotoxicity Syndrome (ICANS)
Description: The Proportion of participants with reported ICANS as defined by the American Society for Transplantation and Cellular Therapy (ASTCT) will be reported
Time Frame: Up to 30 days after discontinuing study treatment, approximately 1 year and 8 months
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Participants Discontinuing Treatment Due to Toxicity
Description: The proportion of participants who reported discontinuing treatment due to a treatment-related toxicity will be reported.
Time Frame: Up to 30 days after discontinuing study treatment, approximately 1 year and 8 months
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 3
proportion of participants | 0

6. Secondary Outcome: Proportion of Participants by Best Achieved Response Rate
Description: The proportion of patients achieving progressive disease, stable disease, partial response, very good partial response, complete response, stringent complete response for best-achieved response, using the IMWG criteria for assessing response, at any time during pembrolizumab therapy will be reported.
Time Frame: Approximately 1 year and 8 months
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Overall Survival (OS) at 12 Months
Description: For OS, participants who remain alive at the end of study follow-up will be censored at the time when the participants is known to be alive. Results will be summarized using the Kaplan-Meier method. The 12-months percentage of participants alive, 25th percentile, median, and 75th percentile, along with corresponding 95% confidence intervals, will be reported.
Time Frame: Up to 2 years
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

8. Secondary Outcome: Median Progression-Free Survival (PFS) at 12 Months
Description: For PFS, participants without progression or death will be censored at the time of the last evaluable disease assessment, while participants without a disease assessment will be censored at the date of first study treatment received. Results will be summarized using the Kaplan-Meier method. The 12-months event-free probabilities, 25th percentile, median, and 75th percentile, along with corresponding 95% confidence intervals, will be reported.
Time Frame: Up to 1 year
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

9. Secondary Outcome: Median Progression-Free Survival (PFS) at 24 Months
Description: For PFS, participants without progression or death will be censored at the time of the last evaluable disease assessment, while participants without a disease assessment will be censored at the date of first study treatment received. Results will be summarized using the Kaplan-Meier method. The 24-months event-free probabilities, 25th percentile, median, and 75th percentile, along with corresponding 95% confidence intervals, will be reported.
Time Frame: Up to 2 years
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

10. Secondary Outcome: Median Duration of Response (DOR)
Description: Median duration of response among the responders will be reported along with 95% confidence intervals.
Time Frame: Up to 2 years
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

11. Secondary Outcome: Cumulative Incidence Function for Time to Next Treatment (TNT)
Description: Competing risks analysis will be performed for analyzing TNT, with death as a competing event. For patients who are alive and do not receive the next line of therapy, TNT will be censored at the last study contact. Cumulative incidence function, along with 95% confidence intervals, will be reported for TNT.
Time Frame: Up to 2 years
Population: Data not collected
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed earlier than expected due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT05191472/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT05191472/ICF_001.pdf